CLINICAL TRIAL: NCT05474248
Title: Effects of A Biofeedback-assisted Diaphragmatic Breathing Training on Postpartum Anxiety: A Randomized Controlled Trial
Brief Title: Diaphragmatic Breathing Training on Postpartum Anxiety
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Ministry of Science and Technology, Taiwan (Other Government)
Collaborators: Taichung Tzu Chi Hospital (Other)
Responsible Party: Principal Investigator, Yuh-Kae Shyu, Assistant Professor, Ministry of Science and Technology, Taiwan
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TCRD-TPE-110-61
Record Dates: First submitted 2022-07-22; First posted 2022-07-26 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Postpartum Anxiety
Keywords: postpartum anxiety; biofeedback; diaphragmatic breathing

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diaphragmatic Breathing Training (Experimental): The experimental group will undergo the diaphragmatic breathing training assisted with StressEraser to breath slowly 4-6 times per minute and practice 15 minutes twice daily.
  Interventions: Behavioral: Experimental group
- Control group (No Intervention): Usual care

INTERVENTIONS:
Behavioral: Experimental group — Diaphragmatic Breathing Training
  Arms: Diaphragmatic Breathing Training

SUMMARY:
This is a two-group pretest-posttest, triple-blinded and randomized controlled trial examining the effects of a biofeedback-assisted diaphragmatic breathing training on postpartum anxiety. This study will include full-term postpartum women, aged from 20 to 49, who experienced anxious symptoms with State Anxiety Inventory (A-State) scored 40 or more at the first postpartum day. Participants will be randomly assigned to either an experimental group (n = 64) or a control group (n = 64). The experimental group will undergo the diaphragmatic breathing training assisted with StressEraser to breath slowly 4-6 times per minute and practice 15 minutes twice daily. Participants in the control condition receive postpartum usual care. The outcome measures include anxiety measured by State-Trait Anxiety Inventory (STAI) and the physiological parameters expressed by blood pressure (BP) and heart rate (HR). Measurements will be taken at the first postpartum day and one month postpartum. We except this breathing training design is able to improve women's postpartum anxiety, and in turn improve their physio-psychological health, breastfeeding and baby care skills.

DETAILED DESCRIPTION:
Ditto

ELIGIBILITY:
Inclusion Criteria:

* full-term postpartum women
* aged from 20 to 49
* STAI-S scored 40 or more at the first postpartum day

Exclusion Criteria:

* newborn with severe illness or stillbirth
* maternal suicide or self-harm
* drug use: sedatives, hypnotics or antipsychotic drugs

Ages: 20 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 128 (Estimated)
Dates: Start 2021-02-28 (Actual); Primary Completion 2021-04-12 (Actual); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Postpartum anxiety | Baseline: postpartum day 1-3
  Assessments using the State-Trait Anxiety Inventory-State (STAI-S) for self-reported anxiety symptoms
Postpartum anxiety | Post-test: Change from baseline postpartum anxiety at 4 weeks postpartum
  Assessments using the State-Trait Anxiety Inventory-State (STAI-S) for self-reported anxiety symptoms

SECONDARY OUTCOMES:
Heart rate | Baseline: postpartum day 1-3
  Assessments using A&D sphygmomanometer (Model 767Plus, A&D Co., LTD., Japan) for heart rate
Heart rate | Post-test: Change from baseline heart rate at 4 weeks postpartum
  Assessments using A&D sphygmomanometer (Model 767Plus, A&D Co., LTD., Japan) for heart rate
Blood pressure | Baseline: postpartum day 1-3
  Assessments using A&D sphygmomanometer (Model 767Plus, A&D Co., LTD., Japan) for systolic blood pressure and diastolic blood pressure
Blood pressure | Post-test: Change from baseline heart rate at 4 weeks postpartum
  Assessments using A&D sphygmomanometer (Model 767Plus, A&D Co., LTD., Japan) for systolic blood pressure and diastolic blood pressure

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Tzu Chi Hospital, Taipei, Xindian Dist, Taiwan